CLINICAL TRIAL: NCT07224490
Title: Kisspeptin to Quantify GnRH Neuronal Function in Health and Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stephanie B. Seminara, MD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 565179; R37HD043341 (NIH)
Record Dates: First submitted 2025-11-03; First posted 2025-11-04 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Reproductive Disorder; Neurodegeneration; SARS-CoV 2
Keywords: Reproductive disorder; Neurodegeneration; SARS-CoV 2; Kisspeptin
MeSH Terms: conditions — Nerve Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Kisspeptin administration (Experimental): Single bolus of kisspeptin
  Interventions: Drug: Kisspeptin 112-121

INTERVENTIONS:
Drug: Kisspeptin 112-121 — Single bolus of kisspeptin
  Other Names: Metastin 45-54

SUMMARY:
The objective of this protocol is to use a case-control paradigm to compare the response to an intravenous administration of kisspeptin in individuals with and without post-covid-19 syndrome. The study subjects will receive a single bolus of kisspeptin.

This study will utilize the technique of frequent blood sampling (q10 minutes) to provide detailed neuroendocrine characterization of endogenous LH secretion before and after kisspeptin administration. This frequency of blood sampling is required to define the features of LH pulses.

DETAILED DESCRIPTION:
Delivery of Interventions:

* 1-2 hours of q10 minute blood sampling
* Administration of a single kisspeptin bolus in a dosing range of 0.313 - 13.19 μg/kg

ELIGIBILITY:
Inclusion Criteria

* Female (ages 18-45 years) or Male (ages 18-60 years)
* Normal blood pressure (systolic BP < 140 mm Hg, diastolic < 90 mm Hg)
* Hemoglobin no less than 0.5 g/dL below the lower limit of the sex specific reference range
* No current or recent use of a medication (including hormonal replacement) that, in the opinion of a study investigator, can modulate the reproductive axis or willing to complete an appropriate washout for that particular medication and its method of administration
* For women, negative serum hCG pregnancy test
* For cases, diagnosis of post-covid-19 syndrome
* For controls, history of prior covid infection but no diagnosis of post-covid-19 syndrome

Exclusion Criteria

* Any condition (medical, mental, or behavioral) that, in the opinion of a study investigator, would likely interfere with participation in/completion of the protocol
* Excessive alcohol consumption (>10 drinks/week)
* Active use of illicit drugs
* For women,
* Pregnant
* Trying to become pregnant during protocol participation
* Breast feeding
* History of any of the following: bilateral oophorectomy (ovaries were removed), breast cancer, thromboembolic disease, coronary artery disease, stroke, thrombophilic disorders, or undiagnosed abnormal genital bleeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Difference in mean luteinizing hormone (LH) amplitude between cases and controls | Day of study visit (one to two hours)
  Difference between cases and controls of mean LH amplitude in response to kisspeptin

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No